CLINICAL TRIAL: NCT04096963
Title: Observe the Safety and Effectiveness of the WATCHMAN FLX™ Left Atrial Appendage Closure (LAAC) Device for Subjects With Non-valvular Atrial Fibrillation to Reduce the Risk of Stroke in Hong Kong Area
Brief Title: Observe the Safety and Effectiveness of the WATCHMAN FLX™ for Subjects in Hong Kong
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2461
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Non-valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- The WATCHMAN FLX Delivery System: Patients who are eligible for a WATCHMAN FLX device according to current international and local guidelines (and future revisions) and per physician discretion;
  Interventions: Device: The WATCHMAN FLX Delivery System

INTERVENTIONS:
Device: The WATCHMAN FLX Delivery System — WATCHMAN FLX Delivery System permit device placement in the LAA via femoral venous access and crossing the inter-atrial septum into the left atrium

SUMMARY:
The primary objective of this study is to observe the safety and effectiveness of the WATCHMAN FLX™ Left Atrial Appendage Closure (LAAC) Device for subjects with non-valvular atrial fibrillation to reduce the risk of stroke in Hong Kong area.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, multi-center observational study. The primary Effectiveness Endpoint is the occurrence of non-effective LAA closure defined as any peri-device flow > 5mm demonstrated by TEE/CT/MRI at First Follow-up.The primary safety endpoint is the occurrence of one of the following events between the time of implant and within 7 days following the procedure or by hospital discharge, whichever is later: all-cause death, ischemic stroke, systemic embolism, or device or procedure related events requiring open cardiac surgery or major endovascular intervention such as pseudoaneurysm repair, AV fistula repair, or other major endovascular repair. Secondary effectiveness endpoint is the occurrence of ischemic stroke or systemic embolism at 12 months from the time of implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are eligible for a WATCHMAN FLX device according to current international and local guidelines (and future revisions) and per physician discretion;
2. Patients who are willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center;
3. Patients whose age is 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility.
2. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion);
3. The subject is unable or not willing to complete follow-up visits and examination for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with non-valvular atrial fibrillation to reduce the risk of stroke
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chan Chin Pang Gary, Principal Investigator — Prince of Wales Hospital; Fung Chi Yan Raymond, Principal Investigator — Princess Margaret Hospital, Canada; Tsui Kin Lam, Principal Investigator — Pamela Youde Nethersole Hospital; Simon Lam, Principal Investigator — Queen Mary Hospital, Hong Kong; SF Chui, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: WATCHMAN FLX HK study completed FPI on 19 Jun 2020, and completed LPI on 8 Oct 2021, took almost 16 months to complete recruiting 50 patients. There are 50 subjects enrolled in study.
Pre-assignment Details: Subjects who meet the eligibility criteria, have signed and dated the Informed Consent Form and actually undergo a WATCHMAN FLX implant procedure are considered enrolled in the study. Baseline data from subjects who meet the eligibility criteria, have signed and dated the Informed Consent Form but do not eventually undergo a WATCHMAN FLX implant procedure are collected for epidemiological reasons, to better characterize the population.
Groups:
- The Subjects Who Complete the Study: Subjects who sign informed consent, meets eligibility criteria and successfully implanted with the WATCHMAN FLX device and complete the study.
Period: Overall Study
Arm/Group | The Subjects Who Complete the Study
Started | 50
Completed | 46
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- The Subjects With No-valvular Atrial Fibrillation Who Implant the WATCHMAN FLX LAAC.: Subjects who meet the eligibility criteria, have signed and dated the Informed Consent Form and actually undergo a WATCHMAN FLX implant procedure.
Arm/Group | The Subjects With No-valvular Atrial Fibrillation Who Implant the WATCHMAN FLX LAAC.
Number analyzed (Participants) | 50
Age, Customized [Mean (Standard Deviation); unit: years]
  Age analysis result | 75 (7.7)
Sex/Gender, Customized [Number; unit: participants]
  Female participants number | 17
  Male participants number | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 50

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint
Description: The occurrence of non-effective LAA closure defined as any peri-device flow > 5mm demonstrated by TEE/CT/MRI at First Follow-up.
Time Frame: First Follow-up (30 ~ 100 days);
Population: A total of 46 participants completed the first follow up and belong to PPS set.
Measure: Number (95% Confidence Interval); unit: percentage of occurence
Groups:
- The Participant Who is PPS Set.: The participant with a completed first follow-up visit is PPS set.
Arm/Group | The Participant Who is PPS Set.
Number analyzed (Participants) | 46
percentage of occurence | 0 [0.0 to 7.7]

2. Primary Outcome: Primary Safety Endpoint
Description: The occurrence of one of the following events between the time of implant and within 7 days following the procedure or by hospital discharge, whichever is later: all-cause death, ischemic stroke, systemic embolism, or device- or procedure-related events requiring open cardiac surgery or major endovascular intervention such as pseudoaneurysm repair, AV fistula repair, or other major endovascular repair. Percutaneous catheter drainage of pericardial effusions, snaring of an embolized device, thrombin injection to treat femoral pseudoaneurysm and nonsurgical treatments of access site complications are excluded from this endpoint.
Time Frame: First Follow-up (30-100 days)
Population: T
Measure: Number (95% Confidence Interval); unit: percentage of occurence
Groups:
- The Subjects With No-valvular Atrial Fibrillation Who Implant the WATCHMAN FLX LAAC.: The subjects with no-valvular atrial fibrillation who implant the WATCHMAN FLX Left Atrial Appendage Closure (LAAC).
Arm/Group | The Subjects With No-valvular Atrial Fibrillation Who Implant the WATCHMAN FLX LAAC.
Number analyzed (Participants) | 50
percentage of occurence | 2.0 [0.1 to 10.6]

3. Secondary Outcome: Secondary Endpoint
Description: The occurrence of ischemic stroke or systemic embolism at 12 months from the time of implant.
Time Frame: 12-Month Follow-up (365 ± 30 days)
Population: A total of 46 participants belong to PPS set and 50 participants belong to ITT set.
Measure: Number; unit: participants
Groups:
- The Participant Who is PPS Set.: The participant who is completed first follow-up visit belongs to PPS set.
- The Participant Who is ITT Set: The subject who enrolled to study.
Arm/Group | The Participant Who is PPS Set. | The Participant Who is ITT Set
Number analyzed (Participants) | 46 | 50
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 0-12months post LAAC.
Groups:
- The Subjects Who Are Attempted or Implanted the WATCHMAN FLX LAAC: The subjects with no-valvular atrial fibrillation who are attempted or implanted the WATCHMAN FLX Left Atrial Appendage Closure (LAAC).
Arm/Group | The Subjects Who Are Attempted or Implanted the WATCHMAN FLX LAAC
All-Cause Mortality (participants affected / at risk) | 3/50
Serious Adverse Events (participants affected / at risk) | 23/50
Other Adverse Events (participants affected / at risk) | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Subjects Who Are Attempted or Implanted the WATCHMAN FLX LAAC (N=50)
Intracranial haemorrhage (Nervous system disorders) | 1 (1)
urinary tract infection (Infections and infestations) | 2 (2)
Pheumonia (Infections and infestations) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Convulsion (Facial & Limb Twitching) (Nervous system disorders) | 1 (1)
General weakness (General disorders) | 1 (1)
Low back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ischemic Stroke (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Fast Atrial Fibrillation (Cardiac disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Right leg involuntary movement (Nervous system disorders) | 1 (1)
Eseherichia coli septicaemia (Infections and infestations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2)
Malignant Urethral tumor (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Right groin wound oozing, postoperative (General disorders) | 1 (1)
Diverticulosis of colon (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Acute decompensated heart failure (ADHF) (Cardiac disorders) | 1 (1)
Bleeding from the HD Catheter Site (General disorders) | 1 (1)
Cardiac Chest Pain (Cardiac disorders) | 1 (2)
Chronic Diarrhea (Gastrointestinal disorders) | 1 (1)
Collapse of lumbar vertebra (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
fever (General disorders) | 2 (2)
Heart Failure (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
INTRACEREBRAL HEMORRHAGE (ICH) (Nervous system disorders) | 1 (1)
Irreducible Left Inguinoscrotal Hernia (Gastrointestinal disorders) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1)
Ischaemic Heart Disease (Cardiac disorders) | 1 (5)
Malignant rectal poylp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
Parotid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Postmenopausal bleeding (Reproductive system and breast disorders) | 1 (1)
right leg swelling (General disorders) | 1 (1)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
ncope (Nervous system disorders) | 1 (1)
Todd's paralysis (Nervous system disorders) | 1 (1)
Wound Hematoma (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Subjects Who Are Attempted or Implanted the WATCHMAN FLX LAAC (N=50)
Dizziness (Nervous system disorders) | 1 (1)
Drug Allergy (Immune system disorders) | 1 (2)
Abrasion wound (Shaving) (Injury, poisoning and procedural complications) | 1 (1)
chest pain of unknown etiology (General disorders) | 1 (1)
COVID-19 infection (Infections and infestations) | 2 (2)
Ischaemic Heart Disease (Cardiac disorders) | 1 (1)
Thrombus (Vascular disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tuberculosis of Lung (Infections and infestations) | 1 (1)
Chronic Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Chalazion (Eye disorders) | 1 (1)
Sprain foot (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT04096963/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT04096963/SAP_001.pdf